CLINICAL TRIAL: NCT01905956
Title: Double-blind, Randomized, Placebo-controlled, Bicentric Clinical Investigation to Evaluate Safety and Efficacy of IQP- AK-102 in Reducing Body Weight in Overweight and Obese Subjects
Brief Title: Safety and Efficacy of IQP- AK-102 in Reducing Body Weight
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: InQpharm Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INQ/010013
Record Dates: First submitted 2013-07-19; First posted 2013-07-23 (Estimated); Results first posted 2016-03-08 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2015-03

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- IQP-AK-102 (Active Comparator): 2 capsules per dose, three times daily
  Interventions: Dietary Supplement: IQP-AK-102
- Placebo (Placebo Comparator): 2 capsules per dose, 3 times daily
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: IQP-AK-102 — IQP-AK-102 was presented in the form of a capsule containing proprietary, patent pending combination of three soluble fibres and excipients.
  Arms: IQP-AK-102
Dietary Supplement: Placebo — The placebo contained microcrystalline cellulose and other excepients. Both active and placebo capsules had identical physical appearance in terms of size, shape, colour and opacity.
  Arms: Placebo

SUMMARY:
The individual ingredients in IQP-AK-102 have been widely used. Backed by data from several studies demonstrating their efficacy, we are conducting this study to look into the efficacy and safety of this novel combination of three fibres, in appetite regulation.

DETAILED DESCRIPTION:
Appetite regulation plays an important role in determining the food intake, which is a complex process influenced by biological, behavioral and environmental stimuli. Satiation (intrameal satiety) is defined as the process of feeling full and subsequently stopping food consumption during eating, it therefore reduces hunger and limits the energy consumptions during meals. On the other hand, satiety or more precisely intermeal satiety, delays the onset and possibly reduces the consumption of the next meal. High viscosity and bulking food components such as dietary fibre are expected to elicit stronger satiation/satiety than macronutrients or clear liquid.

Due to its unique physicochemical properties, dietary fibre has been recognized as a potential ingredient that helps to enhance the sensation of satiety in the upper gut by increasing gastric distension and delaying gastric emptying, which subsequently reduces the food intake, and eventually leading on to weight loss.

The investigational product is formulated from IQP-AK-102, a proprietary, patent pending combination of three soluble fibres. In-vitro studies showed synergistic properties for the fibres in IQP-AK-102. When consumed orally, IQP-AK-102 capsules dissolve in the stomach to release the fibres. Once hydrated, the fibres swell to form a thick, viscous and indigestible gel structure in the stomach. This physical structure results in increased gastric distension and delays the gastric emptying that induces satiety and fullness.

However the unique composition of IQP-AK-102 had not been evaluated in human clinical studies. The objective of this placebo controlled, double blind study was to confirm the benefit of IQP-AK-102 in weight loss through promoting satiety and managing appetite. In this study, 120 overweight and obese subjects (60 per study arm) were tested to investigate if IQP-AK-102 is effective in reducing body weight over a period of 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years
* 25≤BMI≤35
* Expressed desire for weight loss
* Accustomed to 3 main meals/day
* Generally in good health
* Consistent and stable body weight 3 months prior to study enrolment
* Consistent regular physical activity
* Commitment to avoid the use of other weight loss products during study
* Commitment to adhere to diet and lifestyle recommended for the study

Exclusion Criteria:

* Known sensitivity to the ingredients of the device
* Presence of any active gastrointestinal disease
* Malabsorption disorders
* Pancreatitis
* Stenosis in the GI tract
* Bariatric surgery
* Any other reason deemed suitable for exclusion, per investigator's judgement

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2013-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Udo Bongartz, Principal Investigator — analyze & realize GmbH
Locations (1):
- Barbara Grube, Berlin, State of Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- IQP-AK-102: 2 capsules per dose, three times daily
  IQP-AK-102
- Placebo: 2 capsules per dose, 3 times daily
  Placebo
Period: Overall Study
Arm/Group | IQP-AK-102 | Placebo
Started | 60 (Randomized) | 59 (Randomized)
Intention-to-treat Population | 57 (Intention-to-treat population) | 54 (Intention-to-treat population)
Completed | 54 (Per-protocol population) | 48 (Per-protocol population)
Not Completed | 6 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IQP-AK-102 | Placebo | Total
Number analyzed (Participants) | 57 | 54 | 111
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 57 | 54 | 111
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.9 (12.3) | 46.3 (10.5) | 47.4 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 43 | 83
  Male | 17 | 11 | 28
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 57 | 54 | 111
Region of Enrollment [Number; unit: participants]
  Germany | 57 | 54 | 111
Height [Mean (Standard Deviation); unit: centimetres (cm)] | 169.3 (9.6) | 168.2 (9.0) | 168.8 (9.3)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 83.0 (12.4) | 80.8 (8.8) | 81.9 (10.8)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per metre square (kg/m^2)] | 29.3 (2.7) | 29.0 (2.1) | 29.2 (2.4)
Waist Circumference [Mean (Standard Deviation); unit: centimetres (cm)] | 102.1 (10.8) | 98.5 (6.9) | 100.4 (9.2)
Hip Circumference [Mean (Standard Deviation); unit: centimetres (cm)] | 110.2 (8.3) | 108.7 (7.8) | 109.5 (8.1)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 123.9 (9.2) | 128.1 (15.7) | 125.9 (12.9)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 79.7 (6.2) | 81.3 (9.4) | 80.5 (7.9)
Heart Rate [Mean (Standard Deviation); unit: Beats per minute] | 70.6 (5.3) | 70.7 (5.5) | 70.6 (5.4)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Body Weight From Baseline to Week 12
Description: Body weight (kg) was measured in subjects wearing underwear and no shoes using calibrated weighing scales (Tanita BC-420 SMA).
  Results were reported as value at baseline minus value at week-12, ie. amount of weight loss in (kg) (positive values).
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: kilogram (kg)
Arm/Group | IQP-AK-102 | Placebo
Number analyzed (Participants) | 57 | 54
kilogram (kg) | 3.53 (2.28) | 0.14 (1.84)

2. Secondary Outcome: Mean Change in Waist and Hip Circumference (cm) From Baseline to Week 12
Description: Waist circumference (cm) was measured at the level midway between the lateral lower rib margin and the iliac crest.
  Hip circumference (cm) was measured as the maximal circumference over the buttocks.
  Results were reported as value at baseline minus value at week-12, ie. amount of waist and hip circumference reduction (cm) (positive values).
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: centimetre (cm)
Arm/Group | IQP-AK-102 | Placebo
Number analyzed (Participants) | 57 | 54
centimetre (cm)
  Waist Circumference | 2.12 (2.99) | 0.92 (3.24)
  Hip Circumference | 2.25 (2.41) | 1.07 (1.20)

3. Secondary Outcome: Mean Change in Body Fat Content (%) From Baseline to Week 12
Description: Body fat content (%) was measured by bio-impedance method using validated electronic weighing scales (Tanita BC-420 SMA).
  Results were reported as value at baseline minus value at week-12, ie. reduction of body fat content (%) (positive values).
Time Frame: Baseline and 12 weeks
Population: Analysis of body fat was not performed for 1 subject (placebo) due to missing data from Visit 2 - Visit 5. At Visit 1, analysis was performed for 109 subjects only. As such, short of 1 baseline date.
Measure: Mean (Standard Deviation); unit: Percentage of body fat (%)
Arm/Group | IQP-AK-102 | Placebo
Number analyzed (Participants) | 57 | 53
Percentage of body fat (%) | 0.95 (2.91) | 0.08 (1.90)

4. Secondary Outcome: Mean Change in Body Fat Mass (kg) From Baseline to Week 12
Description: Body fat mass kg) was measured by bio-impedance method using validated electronic weighing scales (Tanita BC-420 SMA).
  Results were reported as value at baseline minus value at week-12, ie. reduction of body fat mass kg) (positive values).
Time Frame: Baseline and 12 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: kilogram (kg)
Arm/Group | IQP-AK-102 | Placebo
Number analyzed (Participants) | 57 | 53
kilogram (kg) | 1.32 (2.91) | 0.05 (1.95)

5. Secondary Outcome: Food Craving Questionnaire (FCQ)
Description: This validated questionnaire evaluates changes in food cravings. It contains 15 items and was completed by the subjects based on the momentary feeling at the study site during visits 2 to 5 (Baseline and week 4, 8 and 12). Assessment was based on the following 5-point Likert scale:
  1. = I do not agree at all
  2. = I do not agree
  3. = Neutral
  4. = I agree
  5. = I highly agree
  Results were expressed as the mean score for the whole population in the respective intervention group.
Time Frame: Baseline and 4, 8, and 12 weeks
Population: The analysis is performed for all subjects of the Intention-to-treat population who answered the FCQ at all visits from v2 to v5. Missing data were appeared in 9 cases at visit v5 and additional in 8 cases at visit v4.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | IQP-AK-102 | Placebo
Number analyzed (Participants) | 52 | 47
Units on a scale
  Baseline | 2.65 (1.28) | 2.74 (1.07)
  Week 4 | 2.17 (0.94) | 2.47 (1.04)
  Week 8 | 1.98 (0.96) | 2.34 (0.92)
  Week 12 | 2.31 (1.08) | 2.47 (1.06)

6. Secondary Outcome: Global Evaluation of Efficacy by the Investigators
Time Frame: 12 weeks
Population: The analysis is performed for all subjects of the Intention-to-treat population who answered the questions for the assessment. However, missing data still appeared.
Measure: Number; unit: subjects
Arm/Group | IQP-AK-102 | Placebo
Number analyzed (Participants) | 53 | 45
subjects
  Very Good | 31 | 1
  Good | 18 | 6
  Moderate | 4 | 19
  Poor | 0 | 19

7. Secondary Outcome: Global Evaluation of Efficacy by the Subjects
Time Frame: 12 weeks
Population: as for outcome 6
Measure: Number; unit: subjects
Arm/Group | IQP-AK-102 | Placebo
Number analyzed (Participants) | 54 | 44
subjects
  Very Good | 28 | 1
  Good | 22 | 6
  Moderate | 4 | 22
  Poor | 0 | 15

8. Secondary Outcome: Global Evaluation of Safety by the Investigators
Time Frame: 12 weeks
Population: as for outcome 6
Measure: Number; unit: subjects
Arm/Group | IQP-AK-102 | Placebo
Number analyzed (Participants) | 52 | 43
subjects
  Very Good | 46 | 35
  Good | 6 | 7
  Moderate | 0 | 1
  Poor | 0 | 0

9. Secondary Outcome: Global Evaluation of Safety by the Subjects
Time Frame: 12 weeks
Population: as for outcome 6
Measure: Number; unit: subjects
Arm/Group | IQP-AK-102 | Placebo
Number analyzed (Participants) | 53 | 45
subjects
  Very Good | 46 | 37
  Good | 7 | 7
  Moderate | 0 | 1
  Poor | 0 | 0

ADVERSE EVENTS:
Time Frame: During the treatment period ie. 12 weeks.
Description: The causality of the AEs and intake of IP was assessed by the clinician.
  Three subjects who were excluded (due to violation of inclusion/exclusion criteria, and treatment compliance) in the Intention-to-treat population were included in the adverse events analysis.
Arm/Group | IQP-AK-102 | Placebo
Serious Adverse Events (participants affected / at risk) | 1/58 | 0/56
Other Adverse Events (participants affected / at risk) | 12/58 | 12/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IQP-AK-102 (N=58) | Placebo (N=56)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 — Improbable relation to Investigational product
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IQP-AK-102 (N=58) | Placebo (N=56)
Common cold or upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (4) — Light to moderate
Toothache or dental extraction (General disorders) | 0 (0) | 2 (3)
Gastrointestinal complaints (Gastrointestinal disorders) | 0 (0) | 1 (1)
Headaches and Migraine (General disorders) | 1 (1) | 2 (2)
Distortion and contusion of knee (General disorders) | 1 (1) | 1 (1)
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Abcess of the skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — In the breastbone area
Acute Sciatica (Dorsalgia) (Nervous system disorders) | 0 (0) | 1 (1)
Macular degeneration (Eye disorders) | 0 (0) | 1 (1)
Infection of urinary tract (Renal and urinary disorders) | 0 (0) | 1 (1)
Nausea & Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No